CLINICAL TRIAL: NCT06400537
Title: Clinical Study of Recombinant CD19xCD3 Double Antibody (A-319) in the Treatment of Active/Refractory Systemic Lupus Erythematosus
Brief Title: Clinical Study of A-319 in the Treatment of Active/Refractory Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: ITabMed Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT240243
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; A-319
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A-319 intravenous intervention (Experimental): A-319 will be preset with 3 escalation dose levels by intravenous infusion: dose A, dose B, dose C, total course of treatment: 4 weeks. Anticipated enrollment: 9-18 participants.
  Interventions: Biological: A-319
- A-319 subcutaneous intervention (Experimental): A-319 will be administered via subcutaneous injection at five preset escalating dose levels: Dose A, Dose B, Dose C, Dose D, and Dose E. The total treatment duration is 4 weeks. Each dose group is planned to enroll 3+N (N=0-12) participants, with a total anticipated enrollment of 16-32 study participants.
  Interventions: Biological: A-319

INTERVENTIONS:
Biological: A-319 — A-319 will be dosed according to the assigned group.

SUMMARY:
The purpose of the study is to explore the safety and efficacy of recombinant CD19xCD3 double antibody (A-319) in active/refractory systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
The pathogenic B cells of patients with SLE can produce a large amount of autoantibodies, which will form immune complexes and thereby inducing continuously expanding tissue damage and systemic inflammation. A-319 is a kind of recombinant CD19xCD3 double antibody, it can activate internal T cells to target and kill pathogenic B cells. Clinical trials of A-319 are currently underway in hematological maliganancies concerning B cell abnormality. Preclinical studies have shown the efficacy of A-319 in SLE. The aim of this study is to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity and preliminary efficacy of A-319 in active/refractory SLE. Patients with active/refractory SLE will be invited to participate in the study, to receive A-319 intravenous infusion or subcutaneous injection and follow-up visits of up to 1 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old, regardless of gender;
2. Participants diagnosed with SLE according to the American College of Rheumatology (ACR) 1997 revised criteria for SLE at least 24 weeks prior to signing the informed consent form;
3. Active/refractory systemic lupus erythematosus;
4. Positive test results for at least one of the following autoantibodies at screening: antinuclear antibodies (ANA) immunofluorescence assay at a titer of ≥1:80; anti-dsDNA; or anti-Smith (anti-Sm);
5. Receive the standardized and stable treatment for at least 30 days before the first administration of the study drug;
6. Female participants tested negative for pregnancy, and participants agreed to use effective contraception throughout the trial;
7. Have the ability to understand the nature of the research and voluntarily sign an informed consent form;
8. Participants can communicate well with the researchers and complete all visits according to the requirements of the plan.

Exclusion Criteria:

1. Severe kidney disease;
2. Participants who have central nervous system diseases caused by SLE or non-SLE disease within 8 weeks before the first administration of the study drug;
3. Abnormities of main organ function at screening;
4. Medical history that the researchers believe will pose risk to the safety of the participants, or will affect the safety or effectiveness analysis of the study drug;
5. Active mycobacterium tuberculosis infection;
6. Active hepatitis, or hepatitis B virus surface antigen positive, or hepatitis B virus core antibody positive and hepatitis B virus deoxyribonucleic acid positive, ,or hepatitis C virus (HCV) antibody positive with detectable HCV ribonucleic acid (RNA).;
7. History of human immunodeficiency virus infection, or positive antibodies at screening;
8. Positive syphilis spirochete antibody at screening (except false positive caused by SLE);
9. Participants with chronic active infection or acute infection need systemic anti-infection treatment within 2 weeks before screening, or have superficial skin infection requiring treatment within 1 week before screening;
10. Have undergone major surgery or unhealed wounds, ulcers or fractures within 4 weeks before the first administration of the study drug, or plan to perform major surgery during the study period;
11. Participants diagonosed with malignant tumors within 5 years before screening;
12. History of important organ transplantation or hematopoietic stem cells/or bone marrow transplantation;
13. Have been vaccinated or plan to receive live vaccine or live attenuated vaccine during the research period within 4 weeks before the first administration of the study drug;
14. Participated in any clinical trial within 4 weeks before the first administration of the study drug or within 5 half-lives of the study drug of the clinical trial;
15. Received targeted drugs (rituximab, JAK inhibitors, etc.) at a specific time period before the first administration of the study drug;
16. Received intravenous immunoglobulin, prednisone ≥100mg/d or equivalent glucocorticoid therapy within 4 weeks before the first administration of the study drug, or plasma replacement;
17. Received IL-2, thalidomide, rethidone and traditional Chinese medicine within 4 weeks before the first administration of the study drug;
18. Known allergies to monoclonal antibody drugs, or allergies to A-319 excipients;
19. Participants with depression or suicidal thoughts;
20. Women who are pregnant or breastfeeding, or women who plan to be pregnant or breastfeeding during the study period; or men whose sexual partners plan to become pregnant during the study period;
21. Any reason that the researchers believe will hinder the subject's participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Within 1 year since A-319 infusion
  Safety and tolerability will be assessed by incidence and severity of adverse events (AEs) and serious AEs (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetics of A-319 | Within 1 month since A-319 infusion
  Concentration of A-319 in peripheral blood will be evaluated
Pharmacodynamics of A-319 | Within 1 month since A-319 infusion
  Pharmacodynamics will be assessed by levels of cytokines (IL-6, IL-8, IL-10, IFN-γ, TNF-α) in peripheral blood
Pharmacodynamics of A-319 | Within 1 month since A-319 infusion
  Pharmacodynamics will be assessed by levels of lymphocyte subsets in peripheral blood
Numbers of Participants with positive antidrug antibodies in peripheral blood | Day 28 and month 3 since A-319 infusion
  To evaluate immunogenicity of A-319

OTHER OUTCOMES:
Changes in the Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2000) from baseline | Within 1 year since A-319 infusion (day 15, day 28, month 2, month 3, month 4, month 5, month 6, month 9, month 12)
  Range [0, 105]，higher score represents worse disease activity
Changes in the Physician Global Assessment (PGA) score from baseline | Within 1 year since A-319 infusion (day 15, day 28, month 2, month 3, month 4, month 5, month 6, month 9, month 12)
  Range [0, 3]，higher score represents worse disease activity
Changes in the BILAG-2004 score from baseline | Within 1 year since A-319 infusion (day 15, day 28, month 2, month 3, month 4, month 5, month 6, month 9, month 12)
  Range [0, 72]，higher score represents worse disease activity
Changes in immunological indexes from baseline | Within 1 year since A-319 infusion (day 15, day 28, month 2, month 3, month 4, month 5, month 6, month 9, month 12)
  Serum IgA, IgG, IgE and IgM will be evaluated
Changes in level of anti-nuclear antibody (ANA) in peripheral blood from baseline | Within 1 year since A-319 infusion (day 15, day 28, month 2, month 3, month 4, month 5, month 6, month 9, month 12)
  To evaluate SLE disease activity
Changes in level of anti-double stranded DNA (dsDNA) antibody in peripheral blood from baseline | Within 1 year since A-319 infusion (day 15, day 28, month 2, month 3, month 4, month 5, month 6, month 9, month 12)
  To evaluate SLE disease activity
Changes in levels of complement C3 in peripheral blood from baseline | Within 1 year since A-319 infusion (day 15, day 28, month 2, month 3, month 4, month 5, month 6, month 9, month 12)
  To evaluate SLE disease activity
Changes in levels of complement C4 in peripheral blood from baseline | Within 1 year since A-319 infusion (day 15, day 28, month 2, month 3, month 4, month 5, month 6, month 9, month 12)
  To evaluate SLE disease activity
The therapeutic effect of A-319 on impaired organs in active/refractory SLE patients | Within 1 year since A-319 infusion
  Pathological samples of impaired organs will be analyzed
The clearance effect of A319 on CD19+B cells in active/refractory SLE patients | Within 28 days since A-319 infusion
  To evaluate SLE disease activity
The effect of A-319 on gene expression in peripheral blood lymphocytes of active/refractory SLE | Day 28 and month 3 since A-319 infusion
  To investigate the mechanism of action of A-319 in SLE

CONTACTS AND LOCATIONS:
Overall Officials: Qiubai Li, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Wuhan Union Hospital, Wuhan, Hubei
  - Shanxi Bethune Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No